CLINICAL TRIAL: NCT05177484
Title: An Open Label Randomised Trial to Assess the Efficacy of Post-Operative Ferric Maltol Vs Standard Care for Anaemia Following Colorectal Cancer Surgery
Brief Title: Perioperative Iron for Colorectal Cancer (PICoC Study)
Acronym: PICoC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Royal Wolverhampton Hospitals NHS Trust (Other Government)
Collaborators: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021GAS120
Record Dates: First submitted 2021-11-08; First posted 2022-01-04 (Actual); Results first posted 2025-09-19 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Cancer Colon
MeSH Terms: conditions — Colonic Neoplasms | interventions — ferric maltol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ferric maltol (Experimental)
  Interventions: Drug: oral ferric maltol
- Standard care (No Intervention): Standard post-operative care

INTERVENTIONS:
Drug: oral ferric maltol — The intervention group will commence a course of oral ferric maltol provided oral intake has recommenced and the control group will receive standard care. All patients will have blood tests checked again at day 3 and day 5 postoperatively if they remain as an inpatient. If they are found to be anaemic on either of these two blood tests they will, at this stage, enter their allocated treatment pathway. If a patient shows no evidence of anaemia on either day 2, 3 or 5 blood tests they will be withdrawn from the study. Patients will continue treatment according to their randomisation allocation until 12 weeks after the operation, at which point the patient attends a routine surgical outpatient follow-up clinic. During the outpatient visit the participants will undergo their final blood testing and questionnaire completion.
  Arms: Ferric maltol

SUMMARY:
The PICoC study aims to investigate whether oral ferric maltol given postoperatively offers an improvement in patient and clinician reported outcomes compared to standard care.

DETAILED DESCRIPTION:
Colorectal cancer is associated with iron deficiency anaemia in 40-60% of cases. This anaemia can lead to poorer post-operative outcomes such as higher complication rates, increased length of stay and reduced survival. There has been a recent shift towards the correction of preoperative anaemia in order to optimize perioperative outcomes. However, despite improvements in preoperative haemoglobin there exists a group of patients who develop worsening or recurrent anaemia in the post-operative period. Without intervention up to 90% of patients in the immediate postoperative period may develop anaemia. This is not unexpected given the peri-operative blood loss; poor nutritional intake in the postoperative period; and the frequent blood sampling for laboratory tests. Our data from previous trials has demonstrated that despite preoperative intravenous iron therapy 75% of patients remain anaemic at the time of their colorectal cancer operation. In addition, our unpublished data has found that around 1/3 of patients treated with preoperative iron therapy develop a recurrence of their anaemia in the first year postoperatively. Studies have identified that traditional oral ferrous iron supplementation is largely ineffective for the treatment of postoperative anaemia. However, a newer oral iron preparation - ferric maltol (Ferracru) has been found to be better tolerated and more efficacious than ferrous iron. This study aims to evaluate whether the use of iron supplementation in the form of Feraccru could lead to a more sustained or improved a response in haemoglobin if given after a colorectal cancer operation. Improving this postoperative anaemia may have important implications for clinician and patient reported outcomes. The Perioperative Iron in Colorectal Cancer (PICoC) trial will run as a feasibility study to assess the proposed design, recruitability and outcome measures. Anaemic colorectal cancer patients treated with preoperative intravenous iron will be randomised in an open label design to receive a course of Ferric maltol (intervention group) or standard care (control group) postoperatively. Secondary outcome measures will focus on a comparison of change in blood indices, quality of life, allogenic red blood transfusion rates and postoperative complications between groups. Follow up will continue until the first postoperative outpatient visit at approximately 12 weeks following discharge.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18+ years.
* Diagnosed with histologically or radiologically diagnosed colorectal adenocarcinoma.
* Anaemic at point of diagnosis of colorectal adenocarcinoma (Defined as haemoglobin 10g/L below WHO criteria: 120g/L for males and 110g/L for females, to account for a 10% fluctuation in Hb)
* Undergoing surgery for colorectal cancer with curative intent.
* Date of planned surgery is ≥ 14 days from date of planned initiation of recruitment.
* Able (in the investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Patients who do not have a histological diagnosis of colorectal adenocarcinoma
* Female participants who are pregnant, lactating or planning a pregnancy during the course of the study.
* Patients with evidence of iron overload or disturbances in utilisation of iron as stated in the product SPC.
* Previous gastric, small bowel or colorectal surgery (where ≥50% of stomach or terminal ileum has been resected)
* Chemotherapeutic treatment within the last 4 weeks.
* Known previous anaemia not attributable to colorectal carcinoma (i.e. anaemia in patients with well established, inflammatory disorders)
* Known haematological disease.
* Features necessitating urgent surgery (e.g. obstructive symptoms).
* Previous allergy to intravenous or oral iron or related iron products.
* Patients who are unable to consent.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participants who have participated in another research study involving an investigational product in the past 12 weeks
* Confirmed liver or lung metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2025-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nuha Yassin, Principal Investigator — The Royal Wolverhampton NHS Trust
Locations (1):
- The Royal Wolverhampton NHS Trust, Wolverhampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ferric Maltol | Standard Care
Started | 20 | 20
Completed | 16 | 18
Not Completed | 4 | 2
Not completed — Withdrawn as not anaemic post operatively | 1 | 0
Not completed — Inadvertently withdrawn | 3 | 1
Not completed — Withdrawn as not given standard care, given IV iron | 0 | 1

BASELINE CHARACTERISTICS:
Population: Colorectal cancer patients who were anaemic at diagnosis of their cancer.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferric Maltol | Standard Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Full Range); unit: years] | 74.30 [25 to 93] | 73.5 [49 to 86] | 73.9 [25 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 12 | 12 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White British | 17 | 17 | 34
  Ethnicity: South Asian | 2 | 3 | 5
  Ethnicity: Black British (Caribbean) | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Feasibility of Running the Study, to See if it Could be Run as a Large Multi-centre Study
Description: Feasibility measures will include the number of patients:
  * Eligible from screening
  * excluded and why
  * will stay in the study
Time Frame: 1 year
Population: A total of 42 patients were recruited to the study. There were 2 patients who were withdrawn prior to randomisation. Of those 40 patients randomised 32 patients remained in the study to analysis, this was 80%.
Measure: Number; unit: participants
Arm/Group | Ferric Maltol | Standard Care
Number analyzed (Participants) | 21 | 21
participants | 16 | 18

2. Secondary Outcome: Levels of Haemoglobin and Haematinic Markers (Full Blood Count, Ferritin, Iron, Transferrin, and Transferrin Saturation)
Description: Haemoglobin (Hb) was measured at several timepoints across the study period.
Time Frame: Diagnosis (Baseline), recruitment (at Enrollment), day of surgery (between 2 weeks - 2 months from recruitment), POD2 (2 days post op), POD3 (3 days post op), POD5 (5 days post op), discharge (5 days post op), and follow up (up to 12 weeks)
Measure: Mean (Standard Deviation); unit: g/l
Arm/Group | Ferric Maltol | Standard Care
Number analyzed (Participants) | 16 | 18
g/l
  Hb at Diagnosis | 87 (15.2) | 93.55 (16.01)
  Hb at Recruitment | 106.4 (16.5) | 105 (16.7)
  AHb at Day of Surgery | 116.7 (16.1) | 116.2 (15.9)
  Hb on POD2 | 104.1 (19.6) | 104.0 (12.4)
  Hb on POD3 | 108.8 (16.7) | 106.3 (12.2)
  Hb on POD5 | 103.9 (15.4) | 104.4 (10.46)
  Hb on Discharge | 98.9 (13.4) | 106.2 (10.9)
  Hb Follow Up | 129.7 (19.8) | 128.1 (12.8)

3. Secondary Outcome: Haematinics (Iron Studies)
Description: Iron studies, including total serum iron level, TIBC, transferrin, and transferrin saturation, are essential for diagnosing patients suspected of iron deficiency and overload. Results demonstrated that the Ferric Maltol has improved patents' iron stores.
Time Frame: Recruitment (at Enrollment), day of surgery (between 2 weeks - 2 months from recruitment), POD5 (5 days post op), and follow up (up to 12 weeks)
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Ferric Maltol | Standard Care
Number analyzed (Participants) | 16 | 18
mmol/l
  Iron at recruitment | 8.445 (11.800) | 6.86 (5.790)
  Iron at day of surgery | 13.68 (8.349) | 11.52 (8.900)
  Iron on POD5 | 6.938 (5.302) | 7.328 (4.546)
  Iron follow up | 15.69 (8.931) | 12.97 (6.662)
  Transferrin at recruitment | 3.045 (0.470) | 3.09 (0.740)
  Transferrin at day of surgery | 2.355 (0.397) | 4.265 (7.701)
  Transferrin on POD5 | 1.66 (0.411) | 2.893 (3.028)
  Transferrin follow up | 2.337 (0.4290) | 2.705 (0.553)
  T.Sats at recruitment | 11.49 (15.800) | 9.89 (9.500)
  T.Sats at day of surgery | 23.18 (13.593) | 18.16 (12.303)
  T.Sats on POD5 | 16.46 (11.310) | 15.64 (8.669)
  T.Sats follow up | 26.63 (14.305) | 19.84 (9.846)
  TIBC at recruitment | 75.91 (10.970) | 74.21 (14.140)
  TIBC at day of surgery | 59.11 (9.942) | 62.63 (12.656)
  TIBC on POD5 | 41.68 (10.308) | 47.29 (11.191)
  TIBC follow up | 58.65 (10.769) | 67.81 (13.712)

4. Secondary Outcome: CRP
Description: We looked at the CRP at the different timepoints
Time Frame: Recruitment (at Enrollment), day of surgery (between 2 weeks - 2 months from recruitment), POD2 (2 days post op), POD3 (3 days post op), POD5 (5 days post op), and follow up (up to 12 weeks)
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Ferric Maltol | Standard Care
Number analyzed (Participants) | 16 | 18
mg/dl
  Recruitment | 13.29 (25.65) | 11.8 (13.91)
  Day of surgery | 11.9 (21.30) | 12.55 (14.98)
  POD2 | 137.8 (94.48) | 145.85 (74.62)
  POD3 | 156.8 (101.49) | 136.83 (99.10)
  POD5 | 114.4 (104.32) | 89.6 (94.76)
  Follow up | 4.571 (5.96) | 5.278 (8.46)

5. Secondary Outcome: Side Effects to Ferric Maltol Administration
Description: An aspect of the safety and feasibility of the study was the tolerability of ferric maltol amongst post-operative colorectal cancer patients. We recorded any reported symptoms patient experienced as potential side effects.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Ferric Maltol | Standard Care
Number analyzed (Participants) | 15 | 17
Participants
  No side effects | 10 | 11
  Side effects | 5 | 6

6. Secondary Outcome: Adherence to Treatment
Description: Patients adherence to treatment - if they took their tablets. Both arms are not included as the standard care group did not take Ferric Maltol.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Ferric Maltol
Number analyzed (Participants) | 15
Participants
  All of tablets taken | 11
  Most of tablets taken | 2
  Some of tablets taken | 1
  Few of tablets taken | 1

7. Secondary Outcome: Complications
Description: Differences in rates of complications between the two groups.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Ferric Maltol | Standard Care
Number analyzed (Participants) | 15 | 17
Participants
  Complications | 8 | 9
  No complications | 7 | 8

8. Secondary Outcome: Mortality
Description: Analysis was using Fisher's exact test due to the small sample size, this is approximately 90-day mortality as patients were followed for approximately 12 weeks.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Ferric Maltol | Standard Care
Number analyzed (Participants) | 15 | 16
Participants
  Death | 1 | 0
  Alive | 14 | 16

9. Secondary Outcome: Length of Hospital Stay
Description: Analysing the length of hospital stay of patients in the two groups.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Ferric Maltol | Standard Care
Number analyzed (Participants) | 16 | 18
Days | 7.133 (4.809) | 7.333 (6.202)

10. Secondary Outcome: Readmission
Description: Rates of readmission between the two groups.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Ferric Maltol | Standard Care
Number analyzed (Participants) | 16 | 17
Participants
  Readmission | 2 | 1
  No readmission | 14 | 16

11. Secondary Outcome: Allogenic Blood Transfusion
Description: Patients who required blood transfusion during the trial period.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Ferric Maltol | Standard Care
Number analyzed (Participants) | 4 | 3
Participants
  Pre-operative and intra-operative Transfusion | 3 | 1
  Post-operative Transfusion (During admission) | 1 | 1
  Post-operative Transfusion (Following Discharge) | 0 | 1

12. Secondary Outcome: Grip Strength
Description: Assessed the patients grip strength throughout their perioperative journey.
Time Frame: Recruitment (at Enrollment), day of surgery (between 2 weeks - 2 months from recruitment), POD2 (2 days post op), POD3 (3 days post op), POD5 (5 days post op), and follow up (12 weeks)
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ferric Maltol | Standard Care
Number analyzed (Participants) | 19 | 20
kg
  Recruitment | 23.0868421 (8.49509404) | 23.6342105 (11.4668369)
  Day of Surgery | 23.2763158 (9.41755701) | 24.84 (10.6813364)
  POD2 | 20 (9.21453455) | 21.55 (9.28184502)
  POD3 | 20.2447368 (9.30052111) | 23.01 (10.9261351)
  POD5 | 20.471875 (9.5833183) | 22.2052632 (10.0175526)
  Follow up | 22.7846154 (10.3199117) | 24.2944444 (9.77469556)

ADVERSE EVENTS:
Time Frame: Prior to randomisation, following discharge, during admission, post-operative. Through to study completion, over 19 months
Arm/Group | Ferric Maltol | Standard Care
All-Cause Mortality (participants affected / at risk) | 1/16 | 0/18
Serious Adverse Events (participants affected / at risk) | 6/16 | 4/18
Other Adverse Events (participants affected / at risk) | 4/16 | 3/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferric Maltol (N=16) | Standard Care (N=18)
Hospital stay (Gastrointestinal disorders) | 0 (0) | 1 (1) — Prolonged Hospital Stay for post-operative Ileus, acute kidney injury, supraventricular tachycardia and pneumonia.
Hospital stay (Infections and infestations) | 1 (1) | 0 (0) — Prolonged Hospital Stay with wound infection
Hospital stay (Cardiac disorders) | 0 (0) | 1 (1) — Prolonged hospital stay and unexpected ITU admission with pulmonary embolism and pneumonia
Readmission (Infections and infestations) | 1 (1) | 0 (0) — Readmission for wound infection
Hospital stay (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Prolonged Hospital Stay including treatment for pneumonia.
Hospital stay (Gastrointestinal disorders) | 1 (1) | 0 (0) — Prolonged Hospital stay for post-operative Ileus and acute kidney injury
Readmission (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Readmission and blood transfusion for bleeding per rectum.
Hospital stay (Gastrointestinal disorders) | 1 (1) | 0 (0) — Prolonged Hospital stay for anastomotic bleeding with return to theatre resulting in Ileostomy.
Anastomotic Leak (Gastrointestinal disorders) | 1 (1) | 0 (0) — Anastomotic Leak which resulted in death.
Readmission (Gastrointestinal disorders) | 1 (1) | 0 (0) — Readmission with pain found to have an ischaemic anastomotic stricture.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferric Maltol (N=16) | Standard Care (N=18)
Delirium (Investigations) | 0 (0) | 1 (1) — Delirium following discharged - did not require admission and settled.
Bleed (Surgical and medical procedures) | 1 (1) | 0 (0) — Port site bleed managed conservatively.
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Intermittent Vertigo
Oedema (Surgical and medical procedures) | 1 (1) | 0 (0) — Oedema in lower limbs following surgery. During admission also had a fall with minor head injury and urinary tract infection
Infection (Infections and infestations) | 0 (0) | 1 (1) — Wound infection treated by GP with oral antibiotics.
Side effect of Ferric Maltol (Product Issues) | 1 (1) | 0 (0) — Side effects of Ferric Maltol. Patient reported medication not tolerated due to nausea, diarrhoea, constipation, abdominal pain and headache.
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Rash developed during anaesthetic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT05177484/Prot_SAP_000.pdf